CLINICAL TRIAL: NCT02247817
Title: A Combined Transvenous and Epicardial Lead Placement Procedure for Implantation of Cardiac Resynchronization Devices: a Feasibility Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jasper J. Schouwenburg, Drs., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METc 2013/387
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure With Intraventricular Conduction Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HYBRID (Experimental): Hybrid transvenous/epicardial implantation of a CRT-(D) device.
  Interventions: Device: Hybrid CRT-D/P implantation

INTERVENTIONS:
Device: Hybrid CRT-D/P implantation

SUMMARY:
Cardiac resynchronization therapy has become one of the cornerstones of the treatment of heart failure. However, a large proportion of patients still fails to this type of therapy. This may be due to a suboptimal position of the left ventricular pacing lead, which may be caused by unfavorable cardiac venous anatomy. Implantation of the pacing lead using video assisted thoracic surgery is more flexible and evades the venous system altogether, resulting in a much more favorable position of the pacing lead, with better treatment results as e consequence.

ELIGIBILITY:
Inclusion criteria

* NYHA class II-III.
* Left ventricular ejection fraction ≤ 35%.
* QRS-duration of ≥ 120 ms (NYHA III) or ≥ 130 ms (NYHA II) and left bundle branch block morphology.
* No sidebranch of the coronary sinus near the posterolateral wall of the left ventricle and/or presence of a Thebesian valve which reduces coronary sinus diameter 50% or more (corresponding to a decrease in cross sectional area of 75% or more).
* On optimal medical therapy for heart failure, including beta-blockers, ACE-inhibitors, AT2-antagonists and aldosteron antagonists.
* Age ≥ 18 years.
* Signed informed consent.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Coronary ischemia or a recent myocardial infarction (< 6 months).
* Allready a CRT-device implanted.
* Venous thrombosis without options to reach the right heart.
* Presence of any other condition than HF with a life expectancy of < 1 year.
* History of intrathoracic surgery.
* Presence or suspected presence of a noncompliant left lung.
* Participation in another intervention trial.
* Unable to understand Dutch language.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of procedure related serious adverse events | 30 days after implantation of device